CLINICAL TRIAL: NCT03291262
Title: Survival Outcomes of Ovarian Malignancies in Chinese Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: SOOM-1
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Ovarian Neoplasms; Survival
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Death Domain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow up for death and recurrence — Patients are followed up to determine the specific date of diagnosis, recurrence and death.

SUMMARY:
This study aims to determine survival outcomes (overall survival and progression-free survival) of primary ovarian malignancies in China and relevant risk factors in a prospective cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Primary ovarian malignancies.

Exclusion Criteria:

* Metastatic malignancies to ovaries.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with definite diagnosis of primary ovarian malignancies confirmed by pathologic examinations.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Periods from diagnosis of ovarian cancer to death
Progression-free survival | 5 years
  Periods from diagnosis of ovarian cancer or remission of disease to next recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, China/Beiing, China

REFERENCES:
- [Derived] Sun T, Li L. A cohort study of hypersensitivity reaction in patients with epithelial ovarian cancer treated with carboplatin. Int J Gynecol Cancer. 2019 Mar;29(3):566-571. doi: 10.1136/ijgc-2018-000072. Epub 2018 Dec 22. PMID 30833442